CLINICAL TRIAL: NCT01224977
Title: Development and Validation of a Sputum Biomarker mRNA Panel for the Diagnostic Work-up of Asthma 4.
Acronym: BioSput-Air
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, prof. dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biomarker sputum airway study4
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Asthmatic Patients
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- azithromycin (Other)
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: azithromycin — azithromycin 500 mg 3/week for 3 months

SUMMARY:
The main objectives of the study are:

1. To unravel the importance of molecular phenotyping in predicting the response to antimicrobial therapy with potential anti-inflammatory potency

The investigators have developed a non-invasive technique based on mRNA analysis of induced sputum that enables us to study airway inflammation in detail. This technique forms the basis for our current project based on the following hypotheses:

1. Different molecular asthma phenotypes exist: a Th2 phenotype and a non Th2 phenotype as reported by Woodruff and colleagues (Woodruff PG et al). Sputum mRNA cytokine levels can be used to diagnose Th2 asthma and discriminate this from non-Th2 asthma.
2. Based on our previous research and preliminary data that non-Th2 asthma can be further divided in Th17 asthma and Th1+Th2 asthma; besides these, a fourth group without Th2, Th17 or Th1 characteristics also exist.
3. These subgroups have different responses to anti-microbial therapy with potential anti-inflammatory potency (macrolides).

ELIGIBILITY:
Inclusion Criteria:

* severe asthmatics (GINA step 4 or step 5 (without anti-IgE))

Exclusion Criteria:

* viral/fungal/bacterial infection +fever (<1 month)
* asthma exacerbation (<3 months)
* other respiratory disease (CF, ciliary dyskinesia,bronchiectasis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
sputum cytokine mRNA | 3 months

SECONDARY OUTCOMES:
responsiveness to the medication | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MA Bullens, MD,PhD, Principal Investigator — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België; Sven F Seys, MSc, Study Director — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België
Locations (1):
- University Hospital of Leuven, Leuven, Vlaams-Brabant, Belgium